CLINICAL TRIAL: NCT03558243
Title: Prevention of Radial Artery Occlusion: Comparison of Three HEmostatiC Methods in Transradial Vascular Access for Diagnostic or Therapeutic Coronary Angiography
Brief Title: Prevention of Radial Artery Occlusion: Comparison of Three HEmostatiC Methods in Transradial Intervention
Acronym: PROTHECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart Institute, Mexico (Other Government)
Responsible Party: Principal Investigator, Jesus Reyes, Interventional Cardiology Fellow, National Heart Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PT-18-075
Record Dates: First submitted 2018-05-08; First posted 2018-06-15 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Occlusion of Artery; Radial Artery Injury; Complication
Keywords: radial artery occlusion; prevention; patent hemostasis; transradial intervention; ulnar compression
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The investigator who will evaluate the primary end point will be blinded to which hemostatic technique the patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patent Hemostasis Arm (Active Comparator): The TR Band (Terumo medical) will be placed on the sheath entry site, the air bladder of the TR Band will be filled with 18 mL of air to achieve initial hemostasis. The sheath will be removed, air will be withdrawn slowly until a pulsatile bleeding is observed through the sheath's orifice, once this phenomenon occurs, 2 ml of air will be added to the air bladder and the absence of bleeding will be corroborated, immediately afterwards a pulse oximeter will be placed on the index finger of the patient and transient manual compression of the ipsilateral ulnar artery will be performed, patency of the radial artery will be corroborated by means of oxygen saturation and adequate pulse curve (Barbeau reverse test), if it is not possible to achieve patent hemostasis, it will be retried deflating 1-2 ml of the TR Band every 15 minutes until a positive reverse Barbeau test with absence of bleeding is achieved. TR Band removal will be attempted 2 hours after the procedure.
  Interventions: Procedure: Patent Hemostasis arm
- ULTRA Arm (Experimental): The TR Band will be placed at the sheath entry site, the ipsilateral ulnar artery will be compressed at the Guyon's canal by placing a cylindrical composite made by wrapping 4 inch x 4 inch gauze around a 1-inch plastic needle cap, and compressing it using a circumferentially applied Hemoband. After occlusive compression of ulnar artery is confirmed by means of plethysmography, patent hemostasis protocol will be used for radial artery hemostasis as described at the patent hemostasis arm. The needle cap and hemoband that compresses the ulnar artery will be removed 1 hour after the procedure. TR Band removal will be attempted 2 hours after the procedure.
  Interventions: Procedure: ULTRA arm
- Hemostatic Disc Arm (Experimental): The StatSeal hemostatic disc will be placed above sheath entry site, the TR Band will be placed above the disc, according to the manufacturer's specifications the air bladder will be filled with 8 ml of air, the sheath will be then removed, corroborating the absence of bleeding, 20 minutes later 3 ml of air will be removed, 20 minutes after that 5 ml of air will be removed, finally the investigators will try to remove the deflated TR Band 60 minutes after the procedure.
  Interventions: Device: Hemostatic disc arm

INTERVENTIONS:
Procedure: Patent Hemostasis arm — Patent hemostasis with TR BAND
  Arms: Patent Hemostasis Arm
Procedure: ULTRA arm — Patent hemostasis protocol plus ipsilateral ulnar compression
  Arms: ULTRA Arm
Device: Hemostatic disc arm — StatSeal disc plus TR Band
  Arms: Hemostatic Disc Arm

SUMMARY:
This study evaluates three hemostatic methods for prevention of radial artery occlusion. One third of patients will receive patent hemostasis, another third will receive patent hemostasis plus ulnar compression and the last third will receive the StatSeal hemostatic disc.

DETAILED DESCRIPTION:
The main complication of the transradial access is the occlusion of the radial artery, which although clinically silent in most cases, has been associated with critical hand ischemia, more importantly it limits the radial approach for future coronary interventions, and limits the use of this conduit for coronary revascularization surgery and arteriovenous fistulas.

Factors that prevent occlusion of the radial artery have been identified, including the use of several hemostatic techniques at the conclusion of cardiac catheterization.

The patent hemostasis defined as a technique that allows permeability of the radial artery and at the same time ensures the absence of bleeding was the first hemostatic method that showed a decrease in the incidence of radial artery occlusion, it is currently the quality standard for hemostasis in transradial access worldwide. Recently, the patent hemostasis plus ulnar compression was described, which proved in a randomized clinical trial to be superior to conventional patent haemostasis, decreasing the incidence of radial artery occlusion to 0.8% at 30 days. These hemostatic methods are a subject of current research worldwide. And more clinical trials are expected to confirm the superiority of patent hemostasis plus ulnar compression.

The hemostatic discs used at the beginning as an attempt to reduce the times for the hemostasis of the radial access and therefore the recovery times in units of high volume have attracted attention for their effectiveness and their low incidence of radial artery occlusion, there are few reports who place it as a potential strategy to reduce the incidence of radial artery occlusion. Its effectiveness should be validated in dedicated trials with an adequate sample size.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, both genders, in whom successful transradial access is obtained for elective and urgent diagnostic or therapeutic coronary procedures.

Exclusion Criteria:

* Patients over 18 years of age, both genders, in whom successful transradial access is not achieved and crossover is performed to femoral access.
* Patients over 18 years of age, both genders, who do not give their informed consent to participate in the study.
* Patients over 18 years, both genders, with cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1425 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion (RAO) according to hemostatic technique at 24 hrs and evaluate change at 30 days | 24 Hours and 30 days
  2 Items.
  * RAO at 24 hrs
  * RAO at 30 days
  Measured with Barbeau test.

SECONDARY OUTCOMES:
Vascular Complications | 30 days
  1. 2 items
  * Radial arteriovenous fistula
  * Radial pseudoaneurysm
Hemorrhagic Complications | 24 hours
  1. 2 items
  * Thrombolysis In Myocardial Infarction criteria, Non Coronary Artery Bypass Grafting related bleeding
  * Major bleeding
  * Minor bleeding
  * Minimal bleeding
  * Hematoma formation EASY hematoma scale
  * Grade 1
  * Grade II
  * Grade III
  * Grade IV
  * Grade V
Radial artery occlusion according to heparin dose | 30 days
  1. 3 items
  * RAO with < 5000 Ui heparin dose
  * RAO with 5000-8000 Ui heparin dose
  * RAO with > 8000 heparin dose
Radial artery occlusion according to sheath size | 30 days
  1. 3 items
  * RAO with 5 Fr Sheath's
  * RAO with 6 Fr Sheath's
  * RAO with 7 Fr Sheath´s
Time to TR Band removal | 300 Minutes
  1. 1 Item
  - Averaged time until TR band removal
Radial artery occlusion according to type of procedure | 30 days
  1. 2 items
  * RAO in diagnostic procedures
  * RAO in therapeutic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid-Lidt, MD, Study Director — National Heart Institute, Mexico; Marco A Peña, MD, Study Chair — National Heart Institute, Mexico
Locations (1):
- National Heart Institute, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual patient data will not be shared with other researchers